CLINICAL TRIAL: NCT04355858
Title: Precision Treatment of Luminal Advanced Breast Cancer Based on Molecular Subtyping
Brief Title: Molecularly Targeted Umbrella Study in Luminal Advanced Breast Cancer
Acronym: MULAN
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhimin Shao, Professor, Key Laboratory of Breast Cancer in Shanghai, Department of Breast Surgery, Fudan University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCHBCC-N029
Record Dates: First submitted 2020-04-17; First posted 2020-04-21 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Breast Cancer; Metastatic Cancer
Keywords: first-line therapy
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — famitinib; fluzoparib; pyrotinib; Capecitabine; camrelizumab; Everolimus; Taxes; SHR-1701

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (9):
- NF1 mutated (Experimental): If a patient were NF1 mutated, she would receive SHR7390(MEK1/2 inhibitor) and Faminitib.
  Interventions: Drug: SHR7390; Drug: Famitinib
- gBRCA mutated (Experimental): If a patient were gBRCA mutated, she would receive SHR3162 (PARP inhibitor)and SHR6390(CDK4/6 inhibitor) .
  Interventions: Drug: SHR3162; Drug: SHR6390
- HER2 activated mutated (Experimental): If a patient were HER2 activated mutated and had not previously used capecitabine, she would receive Pyrotinib and Capecitabine , while if the patient have previously used capecitabine, she would only use pyrotinib as a single agent.
  Interventions: Drug: Pyrotinib; Drug: Capecitabine
- PDGFRb mutated (Experimental): If a patient were PDGFRb mutated, she would receive Faminitib.
  Interventions: Drug: Famitinib
- CD8 ≥10% (Experimental): In the arm which IHC showed CD8 ≥10%, this arm will be subdivided into 6 sub-arms, in which Arm 5A-4D, we choose the patients who had CDK4/6 inhibitor before while in Arm 5E, we choose the patients who secondarily resistant to adjuvant endocrine therapy , and in Arm 5FF, we choose the patients who is in stage IV without precious treatment or sensitively recurrence. A patient would receive SHR1210(PD-1 antibody) ,nab-paclitaxel and Faminitib in Arm-5A. A patient would receive SHR1210(PD-1 antibody) and VEGF inhibitor in Arm-5B. A patient would receive SHR1701(PD-L1/TGF-βRII inhibitor) in Arm-5C. A patient would receive SHR1701(PD-L1/TGF-βRII inhibitor) and SHR6390(CDK4/6 inhibitor) in Arm-5D. A patient would receive SHR1210(PD-1 antibody) and SHR6390(CDK4/6 inhibitor) and SERD in Arm-5E. A patient would receive SHR1210(PD-1 antibody) and SHR6390(CDK4/6 inhibitor) and AI in Arm-5F.
  Interventions: Drug: Famitinib; Drug: SHR1210; Drug: Nab paclitaxel; Drug: SHR6390; Drug: SHR1701; Drug: SERD; Drug: AI; Drug: VEGFi
- PAM pathway mutated (Experimental): If a patient had any PAM pathway mutation, she would receive Everolimus(mTOR inhibitor) combined with nab-paclitaxel.
  Interventions: Drug: Everolimus; Drug: Nab paclitaxel
- AR≥10% (Experimental): If a patient's IHC showed AR≥10% , she would receive SHR2554(EZH2 inhibitor) and SHR3680(AR inhibitor).
  Interventions: Drug: SHR2554; Drug: SHR3680
- Epigenetic Cohort (Experimental): In this cohort, a patient would receive SHR2554(EZH2 inhibitor) and SHR3162 (PARP inhibitor).
  Interventions: Drug: SHR3162; Drug: SHR2554
- Combined Immunity Cohort (Experimental): In this cohort, a patient would receive SHR6390(CDK4/6 inhibitor) combined with SHR1701(anti-PD-L1/TGF-βRII bifunctional fusion protein) .
  Interventions: Drug: SHR6390; Drug: SHR1701

INTERVENTIONS:
Drug: SHR7390 — MEK1/2 inhibitor
  Arms: NF1 mutated
Drug: Famitinib — Multi-target tyrosine kinase inhibitor
  Arms: CD8 ≥10%; NF1 mutated; PDGFRb mutated
Drug: SHR3162 — PARP inhibitor
  Arms: Epigenetic Cohort; gBRCA mutated
Drug: Pyrotinib — HER1 / HER2 receptor tyrosine kinase inhibitor
  Arms: HER2 activated mutated
Drug: Capecitabine — In Arm III, if the patient had not previously used capecitabine,she would receive pyrotinib and capecitabine, if the patients have previously used capecitabine, she would only used pyrotinib as a single agent.
  Arms: HER2 activated mutated
Drug: SHR1210 — PD-1 antibody
  Arms: CD8 ≥10%
Drug: Everolimus — mTOR inhibitor
  Arms: PAM pathway mutated
Drug: Nab paclitaxel — Albumin bound paclitaxel
  Arms: CD8 ≥10%; PAM pathway mutated
Drug: SHR2554 — EZH2 inhibitor
  Arms: AR≥10%; Epigenetic Cohort
Drug: SHR3680 — AR inhibitor
  Arms: AR≥10%
Drug: SHR6390 — CDK4/6 inhibitor
  Arms: CD8 ≥10%; Combined Immunity Cohort; gBRCA mutated
Drug: SHR1701 — anti-PD-L1/TGF-βRII bifunctional fusion protein
  Arms: CD8 ≥10%; Combined Immunity Cohort
Drug: SERD — Fulvestrant
  Arms: CD8 ≥10%
Drug: AI — aromatase inhibitor
  Arms: CD8 ≥10%
Drug: VEGFi — Bevacizumab
  Arms: CD8 ≥10%

SUMMARY:
This study is a prospective, single-center, open-label, umbrella-shaped phase II clinical study for patients with HR+/HER2- endocrine-resistant advanced breast cancer.

DETAILED DESCRIPTION:
Seven precision treatment cohorts, which targeting NF1 mutation, gBRCA mutation,HER2 mutation, FDGFRb mutation PAM pathway mutations, CD8 and AR, as long as an epigenetic therapy cohort and a combined immunization cohort were initially set up based on gene expression profiles and molecular pathways. The main purpose is to screen valuable treatment cohorts and prepare for subsequent randomized controlled phase III clinical studies with larger sample size.

ELIGIBILITY:
Inclusion Criteria:

* Females ≥18 years old;
* Histologically confirmed HR + / HER2- invasive breast cancer (specific definition: immunohistochemical detection of ER> 10% tumor cell positive is defined as ER positive, PR> 10% tumor cell positive is defined as PR positive, ER and / or PR Positive is defined as HR positive; HER2 0-1 + or HER2 is ++ but negative followed by FISH detection, no amplification, defined as HER2 negative);
* Locally advanced breast cancer (incapable of radical local treatment) or recurrent metastatic breast cancer;
* Patients with HR+/HER2- advanced breast cancer who were previously treated with CDK4 / 6 inhibitor except for Arm 5E-5F;
* Measurable disease according to Response Evaluation Criteria in Solid Tumors v1.1 (RECIST v1.1)
* Has adequate bone marrow function: absolute neutrophil count > 1.5x10ˆ9 /L; platelet count > 75x10ˆ9 /L, hemoglobin > 9g/dL;
* Has adequate liver function: alanine aminotransferase (ALT) ≤1.5×upper limit of normal (ULN), aspartate aminotransferase (AST) ≤3×ULN, alkaline phosphatase (AKP) ≤3×ULN, total bilirubin (TBIL) ≤ 1.5×ULN.
* Has adequate kidney function: serum creatinine ≤1×ULN.Endogenous creatinine clearance> 50 ml / min (Cockcroft-Gault formula);
* Did not receive radiation, molecular targeted therapy or surgery within 3 weeks before the study began, and has recovered from the acute toxicity of previous treatment (if surgery, the wound has completely healed); no peripheral neuropathy or first degree peripheral neurotoxicity ;
* ECOG score ≤ 2 and life expectancy ≥ 3 months;
* Participants voluntarily joined the study, has signed informed consent before any trial related activities are conducted, has good compliance and has agreed to follow-up.

Exclusion Criteria:

* Treatment with chemotherapy, radiotherapy, immunotherapy or surgery (outpatient clinic surgery excluded)within3 weeks prior to initiation of study treatment(bisphosphonates can be used for bone metastasis);
* Symptomatic, untreated, or actively progressing CNS metastases(glucocorticoids or mannitol needed to control symptoms);
* Significant cardiovascular disease(including congestive heart failure, angina pectoris, myocardial infarction or ventricular arrhythmia in the last 6 months);
* Grade ≥ 1 adverse reactions that are ongoing due to previous treatment. Exceptions to this are hair loss or the investigator's opinion should not be ruled out. Such cases should be clearly documented in the investigator's notes;
* Is pregnant or breast feeding;
* Malignant tumors in the past five years (except cured skin basal cell carcinoma and cervical carcinoma in situ).

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 319 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2023-05-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
ORR | Randomization until the first occurrence of disease progression or death from any cause, which ever occurs first, through the end of study (approximately 5 years)
  The proportion of participants whose best outcome is complete remission or partial remission (according to RECIST1.1)

SECONDARY OUTCOMES:
CBR | Randomization until the first occurrence of disease progression or death from any cause, which ever occurs first, through the end of study (approximately 5 years)
  the percentage of subjects with CR+PR+SD and last more than 24 weeks in all of the evaluable subjects
PFS | Randomization until the first occurrence of disease progression or death from any cause, which ever occurs first, through the end of study (approximately 5 years)
  time to progressive disease (according to RECIST1.1)
OS | Randomization to death from any cause, through the end of study (approximately 5 years)
  time to death due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: Zhi-Ming Shao, Principal Investigator — Fudan University
Locations (1):
- Cancer Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Chen MK. Efficacy of PARP inhibition combined with EZH2 inhibition depends on BRCA mutation status and microenvironment in breast cancer. FEBS J. 2021 May;288(9):2884-2887. doi: 10.1111/febs.15730. Epub 2021 Feb 11. PMID 33570247